CLINICAL TRIAL: NCT06262009
Title: Dynamics of AMR Spread, Persistence and Evolution Between Humans, Animals and Their Environment
Acronym: Dyaspeo
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220101; 2023-A02282-43 (Other: IDRCB)
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Antibiotic Resistant Strain; Transmission, Close-Contact
Keywords: antibiotic resistant transmission; transmission between dog and human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human and dog faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- household: House Members (adults and minors) from 175 households owning a dog
  Interventions: Other: human faecal collection; Other: ancillary study

INTERVENTIONS:
Other: human faecal collection — collecting stools 6 times over a 90 days period and complete a questionnaire at the same times: D1, D7, D15, D30, D60 and D90
Other: ancillary study — interviews and/or ethnographic observations for 50 volunteers

SUMMARY:
Humans in contact with animals such as dog owners, may be at risk of antimicrobial resistance (AMR) acquisition. This is the central issue to be investigated in DYASPEO

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) is a global and multifaceted public health problem. Advanced knowledge on AMR has demonstrated that it not only affects humans but is also widely distributed across animals and the environment. A major cause of the AMR burden refers to the capability of AMR to transmit within and between individuals, including between humans and animals. Leading examples of internationally distributed AMR bacteria are Enterobacterial disseminating resistances to extended-spectrum cephalosporins (ESC-E) and carbapenems (CP-E). Yet, the magnitude and pathways of their cross-sectorial transfers are poorly understood.

There is a great concern that humans in contact with animals be at risk of ESC-E/CP-E acquisition. Whereas an increase in ESC-E carriage in farmers in contact with their food-producing animals was reported, AMR transmission to humans through direct contacts with companion animals has been much less studied. Owing the close relationships between pets and owners, and the fact that 50% of households host a dog or a cat in France, the hypothesis of pet ownership being a risk for humans to acquire ESC-E/CP-E appears strongly relevant. The DYASPEO project will investigate this question through a combination of several approaches from field to laboratory studies, and including epidemiology, ecology, molecular and population genomics, studies on intestinal microbiota, modelling and social sciences.

We hypothesize that the interface between humans and companion animals plays a significant role in the transfer of ESC-E/CP-E. This hypothesis is corroborated (i) by recent data in France showing that antibiotic exposure of companion animals is still increasing contrary to all other animal host (e.g. food-producing animals) and (ii) by a recent study from the consortium demonstrating a high AMR prevalence in dogs getting back home after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child planning to live in the same household as his/her dog during the three months following inclusion.
* Planning to live in the same habitat in the next three months following inclusion (except for holidays).
* Written consent of all adults and of at least one of the two parents for minors under parental authority. A different information note will be elaborated for each age category (6-10 yr-old, 10-15 yr-old and 16-18 yr-old).
* Owning a dog recorded for a surgery at the National Veterinary School

Exclusion Criteria:

* Lack of signed informed consent
* Subject in alternating custody
* Subject under legal protection (guardianship)
* Subject deprived of liberty under judicial constraint
* Subject undergoing psychiatric care
* Lack of affiliation to a social security scheme
* Volunteers who do not speak/write French

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The healthy volunteers (dog owners) will be recruited at a single recruitment centre, which is the National Veterinary School (Maisons-Alfort).
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
generation of a list of priorities for future prevention and control strategies to mitigate antimicrobial resistance (AMR) transmission between companion animals and humans | over the 90 days follow up
  mathematical models combining all the data (epidemiological, bacteriological, genomic, sociological) gathered in the project

SECONDARY OUTCOMES:
Rates of AMR acquisitions in one or several housekeepers | over the 90 days follow up
A list in nature of changes in dog microbiota | over the 90 days follow up
A list in magnitude of changes in dog microbiota | over the 90 days follow up
A list in nature of changes in housekeepers microbiota | over the 90 days follow up
A list in magnitude of changes in housekeepers microbiota | over the 90 days follow up
explore unknown parameters of AMR colonization in dogs under various antibiotic exposures | over the 90 days follow up
the generation of a list of sociological factors and potential at-risk practices relevant in the transmission of AMR from dogs to housekeepers | during semi-directive interviews and/or observational periods

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Madec, PHD, Principal Investigator — ANSES
Locations (1):
- the National Veterinary School Alfort, Maisons-Alfort, France

IPD SHARING:
Plan to Share IPD: Undecided